CLINICAL TRIAL: NCT06291636
Title: Re- Admission Rate Among Survived Patients With Acute Respiratory Failure in Mansoura University Respiratory ICU : One Year Study
Brief Title: Re- Admission Rate Among Survived Patients With Acute Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Tamer Awad, lecturer of chest medicine, Mansoura University
Other Study IDs: R.24.01.2451
Record Dates: First submitted 2024-02-20; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Readmission to the intensive care unit (ICU) results in increased consumption of medical resources and costs, and has been proposed as a marker for quality of care. ICU readmission rates have been estimated at 4 to 14% and different risk factors have been proposed by various studies Readmitted patients mostly carry poor prognosis compared to newly admitted ones, in addition to the bad psychological impact for both patient and his family

DETAILED DESCRIPTION:
Intensive care unit (ICU) is a place where it can provide the comprehensive life-saving care for the critically ill patients. Once the patients recover from the critical illness, the patients should be discharged from ICU to general ward for further management Hospitalizations in the intensive care unit (ICU) deal with the most critical illnesses and consume a significant portion of medical expenses. Readmission to the ICU, either due to the reoccurrence of a previous disease or an unrelated new illness, results in further consumption of cost and medical resources, and has been proposed as a marker for quality of care .

Readmission to the intensive care unit (ICU) results in increased consumption of medical resources and costs, and has been proposed as a marker for quality of care. ICU readmission rates have been estimated at 4 to 14% and different risk factors have been proposed by various studies Readmitted patients mostly carry poor prognosis compared to newly admitted ones, in addition to the bad psychological impact for both patient and his family There is a growing interest in determining the main risk factors related to preventable ICU readmissions as well as in developing predictive tools and alerts to help ICU physicians avoid premature ICU discharges Criteria for ICU admission, discharge, and readmission likely vary dramatically from ICU to ICU and from country to country

Aim of Work:

To study the re- admission rate among survived patients with acute respiratory failure in Mansoura University Respiratory ICU during one year 2023

Study Design:

retrospective study patients and Methods After exclusion of patients with missed data, All consecutive adult (>18 years) and admission to pulmonary critical care unit (PCCU) patients at the Mansoura University Hospital from January 2023 till the end of December 2023 were enrolled in the study

All patients were subjected to:

Demographic data (age and gender), admission severity scoring using acute physiology and chronic health evaluation (APACHE II), type of respiratory failure either hypercapnic respiratory failure type II or hypoxemic respiratory failure type I Glasgow coma scale (GCS), underlying comorbidities including dementia, hypertension, congestive heart failure, stroke, chronic kidney disease, liver cirrhosis, and malignancy, use of steroid, mechanical ventilation (MV) and continuous renal replacement therapy, and organ failure in ICU , time of discharge, cause of ICU readmission were collected A readmission event was recorded if the same patient ID was present in the same year; therefore, the follow-up period was different for each patient enrolled with the longest being 1 year Readmission is considered early if it occurs within 72 h an late after 72 h in the same hospital stay

Statistical analysis:

Data will be analyzed using SPSS (statistical package for social sciences) version 22. Qualitative data will be presented as number and percent, Quantitative data will be tested for normality by Shapiro-Wilk test then described as mean and standard deviation for normally distributed data and median and range for non-normally distributed. The appropriate statistical test will be applied according to data type with the following suggested tests: Chi-Square for categorical variable, Student t test and Mann Whitney test.

Ethical consideration:

Study protocol will be submitted for approval by the institutional research board (IRB), Faculty of Medicine - Mansoura University. The research procedures will be conducted in accordance with the principles of the Declaration of Helsinki. Consent will be obtained from each participant in the study after assuring confidentiality. Patients have the right to withdraw from the study at any point of time during the study without penalty.

ELIGIBILITY:
Inclusion Criteria:

* - Age 18 years or more
* Patient with acute respiratory failure (either type I or type II) who were treated with high flow nasal cannula, non-invasive ventilation or invasive mechanical ventilation
* A readmission event was recorded if the same patient ID was present in the same year; therefore, the follow-up period was different for each patient enrolled
* Readmission is considered early if it occurs within 72 h and late if after 72 h of previous admission in the same hospital.

Exclusion Criteria:

* All patient with missed or incomplete data
* All patients died after first admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with acute respiratory failure (either type I or type II)
Sampling Method: Non-Probability Sample
Enrollment: 994 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-20 (Actual)

PRIMARY OUTCOMES:
Length of hospital and ICU stay and Cause of readmission | 1 year
  From the database of Mansour university hospital registration, we collect the following data about all adult patients (>18 years) with acute respiratory failure and admitted to Mansoura University chest department and its related ICU with at least one readmission from start of January 2023 till the end of December 2023:

CONTACTS AND LOCATIONS:
Locations (1):
- Tamer Awad Elsayed, Al Mansurah, Dakhlia, Egypt